CLINICAL TRIAL: NCT00573235
Title: Epidemiology of Community - Associated Extended-spectrum Beta-lactamases (ESBL) Producing Escherichia Coli
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Yohei Doi, Associate Professor, University of Pittsburgh
Other Study IDs: PRO07090323
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Enterobacteriaceae Infections
Keywords: isolates; infection; E coli isolates
MeSH Terms: conditions — Enterobacteriaceae Infections; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — All samples provided to the investigators are deidentified by the honest broker and will be coded with numbers. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location that only the honest broker has access to. The investigators on this study will keep the samples indefinitely. Samples will be kept in the investigator's laboratory located in Scaife Hall, room 812, 3500 Terrace Street. At no time with the research investigators have access to any patient identifers.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to review patients with E. coli infections at the University of Pittsburgh Medical Center (UPMC) from July 1, 2007 to June 30, 2010 to determine if these infections have arisen in the community rather than in hospitals or nursing homes.

DETAILED DESCRIPTION:
This is chart review at UPMC. There is no human interaction.

ELIGIBILITY:
Inclusion Criteria:

* All patients with E. coli, Klebsiella species and Proteus species infections during the time period of the study will be reviewed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with E. coli, Klebsiella species and Proteus species infections during the time period of the study will be reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Review whether ESBL-producing organisms (E. coli, Klebsiella species and Proteus species) are hospital-acquired, healthcare-associated or community-associated. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yohei Doi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States